CLINICAL TRIAL: NCT03689218
Title: Evidence Generation Related to Stunting Prevention Through Multisectoral Approaches Coupled With Appropriate Complementary Feeding Practices in Pishin, Balochistan
Brief Title: Evidence Generation Related to Stunting Prevention in Balochistan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Trust for Vaccines & Immunization (TVI) (Unknown); Department of Health, Government of Balochistan (Unknown); World Food Program (WFP) (Unknown); Nutrition Cell, Government of Balochistan (Unknown); Youth Organization, Balochistan (Unknown)
Responsible Party: Principal Investigator, Dr Sajid Bashir Soofi, Associate Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Stunting Study Balochistan
Record Dates: First submitted 2018-09-27; First posted 2018-09-28 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Stunting; Low Birth Weight; Anemia in Pregnancy
MeSH Terms: conditions — Growth Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): The control arm will receive routine public and private health services available in the area.
- Intervention (Experimental): Pregnant women in intervention arm will receive 30 sachets of Maamta (Nutritious Food Supplement) during pregnancy and first six months of lactation. Children 6-24 months of age will receive 30 sachets of Wawamum (Lipid-Based Nutrient Supplement) every month during the study.
  Interventions: Dietary Supplement: Maamta (Nutritious Food Supplement); Dietary Supplement: Wawamum (Lipid-Based Nutrient Supplement)

INTERVENTIONS:
Dietary Supplement: Maamta (Nutritious Food Supplement) — Pregnant women will receive 30 sachets of Maamta during pregnancy and first six months of lactation.
  Arms: Intervention
Dietary Supplement: Wawamum (Lipid-Based Nutrient Supplement) — Children 6-24 months will receive 30 sachets of Wawamum every month during the study.
  Arms: Intervention

SUMMARY:
The World Food Programme (WFP) has signed MoU with Planning and Development Department of Balochistan in collaboration with Nutrition Cell and National Programme for Family Planning and Primary Health Care, Balochistan for the prevention of stunting. The project will utilize the window of opportunity (1000 days from conception to 2 years) for addressing stunting in children under-two years. Therefore project will recruit pregnant women during first trimester and newborns who delivered from recruited pregnant women will be followed until the age of 2 years. Children 6-12 months of age will be enrolled and followed until the age of two years. The interventions included nutritional supplements during pregnancy, lactation and for children during 6-24 months of age. The project will be implemented in Lady Health Workers (LHWs) covered areas of districts Pishin and Quetta, Balochistan.

DETAILED DESCRIPTION:
The World Food Programme (WFP) has signed MoU with Planning and Development Department of Balochistan in collaboration with Nutrition Cell and National Programme for Family Planning and Primary Health Care, Balochistan for the prevention of stunting. The Stunting Prevention interventions will contribute to revert the trends of chronic malnutrition among children less than 5 years of age. The intervention is coupled with plans to document the impact through credible evidence generation in collaboration with academic institute/s through a research based study in Pishin and Quetta Districts.

Balochistan is the most underdeveloped areas of Pakistan with a very poor health and nutrition situation. According to the National Nutrition Survey (NNS) 2011, the prevalence of stunting in Balochistan is 52% amongst the highest rates in the country. The prevalence of wasting in Balochistan is 16%, indicating a public health emergency. Women and children also suffer from some of the world's highest levels of vitamin and mineral deficiencies with maternal anaemia at 47% in Balochistan and Vitamin A deficiency in children at 74% in Balochistan.

Although a number of nutrition approaches and actions have been implemented in Pakistan at various times, there hasn't been a comprehensive approach to prevent under nutrition in general, and stunting specifically. WFP & MOH will be implementing the nutrition interventions, and this proposal is widely implemented/evaluated in Pakistan, so the project aims to contribute towards to fill the evidence gap for the prevention of stunting through multisectoral approaches coupled with appropriate complementary practices in Balochistan. The evidence base for undernutrition and stunting prevention globally is actually quite well established. There is existent evidence that points to the need to intervene during gestation and the first two years of life (1000 days) to prevent child undernutrition and its consequences. It suggests that investments in interventions during this window of opportunity are likely to have the greatest benefits.

The effectiveness of the project will be measured in terms of the impact of the proposed interventions on the stunting and nutritional outcomes in the target group (children and PLW). Given the conditions of project implementation, a mixed-methods study design including formative research, cross-sectional baseline & endline surveys, cluster randomized controlled trial (RCT) and process evaluation would be appropriate to assess the impact of the intervention. The control clusters will receive routine public and private health services available in the area. The RCT will utilize the window of opportunity (1000 days from conception to 2 years) for addressing stunting in children under-two years. A cohort of children between the age of 6-12 month will also be enrolled in the study and will be followed up to the age of 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women during 1-3 months of pregnancy
* Child age between 6-12 month at the time of enrollment
* Willing to participate in the study and provide informed consent
* Living in catchment area of LHW

Exclusion Criteria:

* More than 4 months of pregnancy
* More than 12 months of child age
* Not willing to participate in the study and unable provide informed consent
* Not living in catchment area of LHW

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2180 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Reduction in stunting in children at 24 months of age | 32 months
  10% reduction in stunting

SECONDARY OUTCOMES:
Improvement in anemia during pregnancy | 9 months
  Improvement in anemia during pregnancy
Improvement in anemia in children | 18 months
  Improvement in anemia in children
Reduction in low birth weight | 9 months
  Reduction in low birth weight in newborns

CONTACTS AND LOCATIONS:
Overall Officials: Sajid B Soofi, FCPS, MBBS, Principal Investigator — Aga Khan University
Locations (2):
- Pakistan (2):
  - District Pishin & Quetta, Quetta, Balochistan
  - Aga Khan University, Karachi, Sindh